CLINICAL TRIAL: NCT01933620
Title: Studies of the Human Microbiome in Clinical Center Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 130180; 13-CC-0180
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-06-26

CONDITIONS: Multidrug-resistant Colonization
Keywords: Multidrug-Resistant Organism; Nosocomial Infection; Natural History
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patients who might become colonized or infected with a multidrug-resistant organism

SUMMARY:
Background:

- The intestines, mouth, and skin all contain billions of bacteria and some fungi. Every person s body contains microorganisms like these. They normally do not make people sick. Researchers are interested in how these microorganisms change when a person is hospitalized. They want to find out if changes take place because of the hospitalization (such as treatments used or changes in medical condition) or because of a person s biology (such as their immune system).

Objectives:

- To understand which microorganisms are most likely to spread through hospitals and what affects that spread.

Eligibility:

- People 2 years of age and older who are going to be inpatients at the National Institutes of Health Clinical Center (NIHCC) for at least 48 hours.

Design:

* Clinicians will take samples from participants up to once a day for as long as they are hospitalized at NIHCC.
* Samples will be taken with a swab, from the rectal area, groin, throat, and armpit, and possibly other areas.
* Participants may give a stool sample or be asked to spit into a cup.
* Clinicians will collect some information from participants medical records. They may request some samples of tissue that are left over from procedures already scheduled at NIHCC.
* After participants leave the NIHCC, samples may be taken when they return for follow-up visits from their hospitalization, for up to 2 years. They will not have to return as a follow-up for this study only....

DETAILED DESCRIPTION:
The goal of this protocol is to explore changes to microbial communities during the course of hospitalcare, and to determine the extent to which these alterations affect whether hospitalized patients become colonized with healthcare-associated organisms. The study enables collection of clinical specimens and associated medical data to evaluate the natural history, epidemiology, and genomics of patients who might become colonized or infected with a multidrug-resistant organism. Biological specimens including stool, sputum, and swabs will be taken from Clinical Center inpatients at least 2 years of age as frequently as daily through discharge, and at follow-up visits for up to 2 years from the date of enrollment. To understand possible pathogen colonization and infection of hospitalized patients, this protocol will assess the full complement of the microbial-host-environmental contributions including: (1) microbial genome and community;(2) patient s genotype, underlying medical condition, medical treatment; and (3) hospital practices and environment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet the following inclusion criteria to participate in the study:

* Be inpatients in the NIH CC with an expected hospitalization of at least 48 hours beyond the date of referral.
* Be 2 years of age or older
* Allow storage of tissue samples for future analyses.
* Allow genetic testing of body fluids, and tissue specimens.

EXCLUSION CRITERIA:

A patient will not be eligible if he/she has any condition which, in the investigator s opinion, places the patient at undue risk by participating in the study.

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals hospitalized at the Clinical Center
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-01-28 (Actual); Primary Completion 2028-10-16 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to accumulate a sufficiently robust body of intestinal microbiome data and clinical and epidemiological metadata to characterize fully the changes in the human microbiota that occur during the course of hospitalization an... | At completion of study
  Once sufficient microbiome data and clinical and epidemiological meta data is collected we will be able to fully characterize the changes in the human microbiota that occur during the course if hospitalization

SECONDARY OUTCOMES:
Determine the features of microbiota that may render patients vulnerable to or protect patients from colonization with MDROs. | At completion of study
Determine clinical correlates of MDRO colonization and infection | At completion of study
Detect the presence of MDROs in biological samples obtained from participants. | At completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Alison Han, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-CC-0180.html